CLINICAL TRIAL: NCT04669795
Title: Evaluation of Osteogenic Potential of Cissus Quadrangularis on Mandibular Alveolar Ridge Distraction
Brief Title: Osteogenic Potential of Cissus Quadrangularis Alveolar Ridge Distraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa Altaweel, Principle Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Al-AlAzhar University
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Distraction of Bone; Dental Implant
Keywords: Alveolar; Bone; Distraction
MeSH Terms: conditions — Diastasis, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): Placebo was given to ten patients during consolidation period ( 2 capsule daily for 6 months during consolidation period)
  Interventions: Drug: Cissus Quadrangularis
- Group 2 (Experimental): Cissus quadrangularis in form of capsules given to ten patients ( 2 capsule daily for 6 months during consolidation period)
  Interventions: Drug: Cissus Quadrangularis

INTERVENTIONS:
Drug: Cissus Quadrangularis — Drug with osteogenic potential given to the patients after consolidation period. dose was two capsules once /day with meals for 6 weeks
  Other Names: Hadiod capsule

SUMMARY:
Deficient alveolar mandibular ridge corrected distraction osteogenesis to facilitate dental implant placement. Patients grouped into 2 groups: one group received Cissus quadrangularis during the consolidation period, and the other group received placebo.

DETAILED DESCRIPTION:
OPGs were taken immediately after distractor placement, at end of activation period, at 1st,2nd month of consolidation period, and at end of consolidation period. Change in bone height was evaluated immediately after distractor placement, at end of activation and end of consolidation periods.

CBCT were taken immediately after implant installation, and 6 months later to evaluate change bone density and marginal bone level about the dental implant.

histological evaluation was done by biopsy obtained, by trephine bur, from implant site during its preparation. The bone biopsy fixed in 4% formalin solution for 7 days, rinsed in water, and dehydrated in sequent phases of ethanol (70, 80, 90, and 100%) and then specimens were stained by hematoxylin- eosin for microscopic evaluation.

Radiographic evaluation

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they were free from any disease that may affect healing. Also, presented with 2-3 missing teeth at least in posterior area and CBCT showed bone height above inferior alveolar canal (IAC) ranged 8-10mm.

Exclusion Criteria:

* patients were excluded if they suffered from any disease affect tissue healing, bad oral hygiene or heavy smoking patients

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Bone gain after distraction | immediately at end of distractor activation
  Increase in bone height after distraction
Relapse after distraction | 3 months from beginning of consolidation period
  Relapse evaluated on panorama
Crestal bone loss around dental implant | 6 months from implant placement
  By using cone beam CT, crestal bone level around implant evaluated by measuring a distance from implant apex to a point on dental implant where bone contacts the dental implant mesially and distally. then average of bone loss round each implant was obtained.
Bone density around dental implant | 6 months from implant placement
  By using cone beam CT, bone density assessed around dental implant at crestal, middle, and apical portions then average was obtained

CONTACTS AND LOCATIONS:
Overall Officials: Altaweel, Principal Investigator — Al-Alharby university
Locations (1):
- Faculty of dental medicine, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altaweel AA, Baiomy AABA, Shoshan HS, Abbas H, Abdel-Hafiz AA, Gaber AE, Zewail AA, Elshiekh MAM. Evaluation of osteogenic potential of Cissus quadrangularis on mandibular alveolar ridge distraction. BMC Oral Health. 2021 Oct 4;21(1):491. doi: 10.1186/s12903-021-01847-y. PMID 34607598